CLINICAL TRIAL: NCT05996913
Title: An Intervention for Somatic Flashbacks in Post-Traumatic Stress Disorder: a Feasibility Study
Brief Title: Feasibility of an Intervention for Somatic Flashbacks in PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Camden and Islington NHS Trust (Other Government); Central and North West London NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 157653
Record Dates: First submitted 2023-07-25; First posted 2023-08-18 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Imagery rescripting intervention for somatic flashback
  Interventions: Other: Imagery rescripting

INTERVENTIONS:
Other: Imagery rescripting — The current project aims to explore the feasibility of intervention featuring imagery rescripting (ImRs) and grounding in the management of somatic flashbacks amongst this population. ImRs was developed as a method to help activate a traumatic memory, bring corrective information into the memory, create a more favourable outcome to the memory and to support the participant to discover and express inhibited trauma-related emotional responses (Arntz & Weertman, 1999).

SUMMARY:
This trial will explore the feasibility and acceptability of an intervention for Somatic flashbacks in Post-Traumatic Stress Disorder (PTSD). Imagery Rescripting (ImRs) will form a central part of the intervention.

The primary objective of this trial is to explore the acceptability and feasibility of delivering an intervention for the management of somatic flashbacks to a population of adults experiencing post-traumatic stress disorder.

The secondary objectives of this trial will be to examine if the intervention leads to any differences in participants experience of somatic flashbacks and their global symptoms of PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a reaction to a traumatic event where a person perceived a high risk of danger to themselves or others (e.g. sexual assault, car crash). Re-experiencing symptoms are a core component to diagnosis and can be understood as intrusive memories of a past traumatic event which are re-experienced involuntarily, as if they are happening in the present and contain more sensory details than nontraumatic memories. These 'intrusive memories' can be experienced as visual, auditory, olfactory, gustatory, and tactile. Other symptoms of PTSD include hyperarousal, emotional numbing and avoidance of stimuli which remind a person of the trauma. Trauma-focussed therapies have an established evidence-base and are widely used to treat PTSD. Their broad aim is to process the memories of a trauma and the meanings attached to it.

The current project seeks to explore the phenomenon of somatic re-experiencing, which we will refer to as somatic flashbacks. Within the field of trauma-focused therapy and research, the experience of somatic flashbacks is acknowledged anecdotally but lacks specific research. The limited research that does exist in this area is descriptive and focuses on somatic flashbacks of pain (see below). There is no existing empirical research exploring the management of somatic flashbacks more generally (e.g. re-experiencing of specific, bodily sensations that were present at the time of the trauma, including internal or external sensations, experience of warmth or coldness, and other physical sensations).

Four existing case reports describe participants who report experiencing somatic flashbacks (of pain) that resemble, in quality and location, the sensations experienced during the traumatic event. This includes: two participants who report waking during surgery; a veteran who re-experienced "pain like a shrapnel wound"; a veteran who re-experienced headaches after losing an eye; and a survivor of the 2005 London bombings who re-experienced pain flashbacks "similar in quality to the original electrocution pain" experienced during the explosion.

An additional study completed over a two-year period to assess the prevalence of pain flashbacks in a sample of participants with PTSD accessing an NHS trauma service reported that 49% of the sample reported experiencing somatic flashbacks of pain.

The current project aims to explore the feasibility of intervention featuring imagery rescripting (ImRs) and grounding in the management of somatic flashbacks amongst this population. ImRs was developed as a method to help activate a traumatic memory, bring corrective information into the memory, create a more favourable outcome to the memory and to support the participant to discover and express inhibited trauma-related emotional responses.

In early studies, various versions of ImRs were used to target symptoms of PTSD. Over the last 30 years, subsequent studies have demonstrated the efficacy of ImRs amongst participants with PTSD who have been injured at work; refugee populations; participants who feel contaminated following childhood sexual abuse; veterans; participants who have experienced childhood trauma; and participants who feel guilt after surviving a traumatic event.

The current project aims to contribute to the existing evidence-base for ImRs in PTSD. It will address the gap in knowledge around the feasibility of ImRs in the treatment and management of somatic flashbacks in PTSD. It will employ a similar intervention used in a pilot study for feelings of shame. The intervention will be developed with the support of experts in the field. They will provide input on the treatment protocol and review intervention recordings to ensure fidelity to the approach.

At the time of writing, no existing studies have explored the use of an intervention featuring ImRs to manage somatic flashbacks in PTSD. Given the lack of existing research, an acceptability and feasibility research design will be employed.

ELIGIBILITY:
Inclusion criteria

* Aged 18 and above
* DSM-5 diagnosis of PTSD or Complex PTSD
* Participants who are currently experiencing somatic flashbacks
* Willing and able to provide written informed consent to treatment

Exclusion criteria:

* Currently receiving another trauma-focussed intervention
* Active suicidal intent or recent (past 8 weeks) suicide attempt
* Currently abusing substances
* Participants whose participation in the study is not considered in their best interest by the clinical team at Traumatic Stress Clinic and Woodfield Trauma Service
* Participants who do not consent to the intervention sessions being recorded
* Participants who do not consent to their assessment information being made available to the trainee clinical psychologist carrying out the intervention

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability/Adherence Scale score | Through study completion, an average of 8 weeks
  The Treatment Acceptability/Adherence Scale measures a participants experience of an intervention. The questionnaire is made of up 10 items and each item is measured on a scale from 1 (disagree strongly) to 7 (Agree strongly).
What percentage of participants using the service are eligible agreed to take part? | 1 year
  The percentage of participants who access the service who meet the eligibility criteria for the intervention
What percentage of participants who are eligible to take part, accept the intervention offer? | 1 year
  The percentage of participants who meet the eligibility criteria for the intervention and agree to take part in the trial.
What percentage of participants completed treatment? | 1 year
  The percentage of participants who agree to take part in the trial who go on to complete the intervention.

SECONDARY OUTCOMES:
Changes in the frequency of somatic flashbacks | Through study completion, an average of 8 weeks
  A visual analogue scale from 0 (not frequent at all) to 100 (extremely frequent)
Changes in the intensity of somatic flashbacks | Through study completion, an average of 8 weeks
  A visual analogue scale from 0 (not intense at all) to 100 (extremely intense)
Changes in the distress associated with somatic flashbacks | Through study completion, an average of 8 weeks
  A visual analogue scale from 0 (not distressing at all) to 100 (extremely distressing)
Changes in participants sense of ability to cope with the somatic flashbacks | Through study completion, an average of 8 weeks
  A visual analogue scale from 0 (not coping at all) to 100 (coping very well)
Changes in global symptoms of PTSD | Through study completion, an average of 8 weeks
  Measured using the PCL-5 questionnaire, which is a 20-item measure. Each item measured on a scale from 0 (not at all) to 4 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Livia Ottisova, Doctorate, Principal Investigator — Camden and Islington NHS
Locations (2):
- United Kingdom (2):
  - Traumatic Stress clinic, London
  - Woodfield Trauma service, London

IPD SHARING:
Plan to Share IPD: No